CLINICAL TRIAL: NCT00371644
Title: Manualized Treatment for Veterans With Military Sexual Trauma
Brief Title: Treatment for Veterans With Military Sexual Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4445-R; IRB 06-036 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Symptoms; Anxiety Symptoms; Quality of Life
Keywords: Stress Disorders, Post-Traumatic; Cognitive Processing Therapy; Military sexual trauma; Psychology, Military; Veterans; Rape; Veterans, psychology; Healthcare utilization
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Military Sexual Trauma | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Participants receive 12 biweekly sessions of Cognitive Processing Therapy (CPT).
  Interventions: Behavioral: Cognitive Processing Therapy
- Arm 2 (Active Comparator): Participants receive 12 biweekly sessions of Present Centered Therapy (PCT).
  Interventions: Behavioral: Present-Centered Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the rape.
  Other Names: CPT
  Arms: Arm 1
Behavioral: Present-Centered Therapy — PCT consists of general support and education focused on current issues in the patient's life. It emphasizes the focus on the individual's current life, and conceptualizes the problems addressed as manifestations of PTSD that, in some cases, may have been present for long periods of time. Emphasis is on problem solving and improving relationships. Connections are made between current problems and PTSD symptoms. PCT provides the emotional support for the trauma patient that is thought to help in recovery and helps the victim gain a better understanding of the nature of the patient's problems and connection with PTSD.
  Other Names: PCT
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Cognitive Processing Therapy (CPT) versus Present-Centered Therapy (PCT) in treating current post-traumatic stress symptoms associated with sexual assault that occurred while veterans were serving in the military.

DETAILED DESCRIPTION:
This study is designed to provide insight into effective treatment of veterans with current Post Traumatic Stress Disorder [PTSD] that resulted from sexual assault that occurred during their active military duty [MST]. This issue is of critical importance, as (1) Congress mandated VA to provide counseling to veterans with sexual trauma. (2) Based on the national MST surveillance data of 1.7 million VA patients, 22% of women and 1% of men have experienced MST. (3) With 20,000 Operation Iraqi Freedom [OIF] veterans having already sought healthcare since deployment, VA will begin to serve a higher percentage of women from combat zones, where the epidemiology of sexual assault and the efficacy of conventional treatments are essentially unknown. Finally, (4) findings from our MST-Study of 270 women veterans strongly suggests that MST is clinically different from civilian adult or child sexual trauma, bringing into question whether conventional civilian-based treatment will be effective with MST veterans.

Cognitive Processing Therapy (CPT) is a therapy developed to treat civilian rape-related PTSD. The efficacy of CPT has been shown with female civilians with sexual assault histories. However, there has not been any research examining the effectiveness of CPT in treating symptoms associated with sexual assault that occurs in military settings. The difference clinically between sexual assault in civilian and military settings is important, as revealed by our clinical experience and empirical findings. In working with veterans with MST for over 13 years we have noted that the assaults are often perpetrated by trusted military personnel and the victim is often without access to immediate treatment or care. Empirically, our research demonstrates that MST is associated with higher rates of PTSD compared to civilian sexual assault.

The primary goal of the study is to evaluate the effectiveness of CPT treatment versus Present Centered Therapy (PCT) for PTSD and associated symptoms resulting from MST. The study objectives will be met by three levels of hypotheses. Hypotheses focus on the primary outcome (PTSD symptoms), confirmatory outcomes (depression symptoms, quality of life), and exploratory outcomes (cost and utilization). Based on the results of the study, we intend to produce an educational CD-ROM, which will include a training manual to educate practitioners on the use of the more effective treatment with veterans. It will be designed for administration by clinicians who represent a range of disciplines (e.g., psychologists, nurses, social workers) and levels of training (e.g., bachelor through doctoral degrees).

This is a randomized controlled clinical trial involving veterans from the VA North Texas Healthcare System (VANTHCS). Data will be obtained from face-to-face interview and written questionnaires at baseline, treatment completion, 2-month, 4-month, and 6-month follow-ups. Patients will be randomized to one of two conditions (CPT or PCT). Patients will receive biweekly sessions of the respective individual therapy from trained therapists for a 6-week period (total of 12 sessions), followed by scheduled assessments. The primary endpoint is the CAPS score, a measure of PTSD severity. Secondary endpoints include anxiety, depression, quality of life, and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Veteran (female or male) from any era with a current diagnosis of PTSD due to MST
* Experienced MST no less than 3 months prior to entering the trial
* Identify that MST is the trauma that is causing the worst current distress (if other traumas also experienced)
* Have at least one clear memory of the trauma (sufficient to write impact statement)
* Consent to be randomized into treatment
* Not receive other psychotherapy during the 6 weeks of active treatment
* (if on psychoactive medications) if new antidepressant, be on stable medication regimen for a minimum of 6 weeks prior to entering the trial (if recent changes to antidepressant dosage or additions or changes of antipsychotic or anti-anxiety medication, eligible immediately)

Exclusion Criteria:

* Current substance dependence
* Prior substance dependence that has not been in remission for at least 3 months
* Any current psychotic symptoms
* Current mania or unstable Bipolar Disorder
* Prominent current suicidal or homicidal features
* Any severe cognitive impairment or history of Organic Mental Disorder
* Current involvement in a violent relationship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alina M Suris, PhD, Principal Investigator — VA North Texas Health Care System, Dallas
Locations (1):
- VA North Texas Health Care System, Dallas, Dallas, Texas, United States

REFERENCES:
- [Result] Suris A, Link-Malcolm J, Chard K, Ahn C, North C. A randomized clinical trial of cognitive processing therapy for veterans with PTSD related to military sexual trauma. J Trauma Stress. 2013 Feb;26(1):28-37. doi: 10.1002/jts.21765. Epub 2013 Jan 16. PMID 23325750
- [Result] Holliday R, Link-Malcolm J, Morris EE, Suris A. Effects of cognitive processing therapy on PTSD-related negative cognitions in veterans with military sexual trauma. Mil Med. 2014 Oct;179(10):1077-82. doi: 10.7205/MILMED-D-13-00309. PMID 25269124
- [Result] Mullen K, Holliday R, Morris E, Raja A, Suris A. Cognitive processing therapy for male veterans with military sexual trauma-related posttraumatic stress disorder. J Anxiety Disord. 2014 Dec;28(8):761-4. doi: 10.1016/j.janxdis.2014.09.004. Epub 2014 Sep 21. PMID 25260214
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Holliday R, Holder N, Monteith LL, Suris A. Decreases in Suicide Cognitions After Cognitive Processing Therapy Among Veterans With Posttraumatic Stress Disorder Due to Military Sexual Trauma: A Preliminary Examination. J Nerv Ment Dis. 2018 Jul;206(7):575-578. doi: 10.1097/NMD.0000000000000840. PMID 29905663
- [Derived] Wiblin J, Holder N, Holliday R, Suris A. Predictors of Unbearability, Unlovability, and Unsolvability in Veterans With Military-Sexual-Trauma-Related Posttraumatic Stress Disorder. J Interpers Violence. 2021 Apr;36(7-8):3814-3830. doi: 10.1177/0886260518777554. Epub 2018 May 31. PMID 29848187
- [Derived] Holliday R, Holder N, Suris A. Reductions in self-blame cognitions predict PTSD improvements with cognitive processing therapy for military sexual trauma-related PTSD. Psychiatry Res. 2018 May;263:181-184. doi: 10.1016/j.psychres.2018.03.007. Epub 2018 Mar 14. PMID 29573657
- [Derived] Holliday RP, Holder ND, Williamson MLC, Suris A. Therapeutic response to Cognitive Processing Therapy in White and Black female veterans with military sexual trauma-related PTSD. Cogn Behav Ther. 2017 Sep;46(5):432-446. doi: 10.1080/16506073.2017.1312511. Epub 2017 May 9. PMID 28485687
- [Derived] Williams R, Holliday R, Clem M, Anderson E, Morris EE, Suris A. Borderline Personality Disorder and Military Sexual Trauma: Analysis of Previous Traumatization and Current Psychiatric Presentation. J Interpers Violence. 2017 Aug;32(15):2223-2236. doi: 10.1177/0886260515596149. Epub 2015 Jul 21. PMID 26198645

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Processing Therapy (CPT): Participants receive 12 biweekly sessions of Cognitive Processing Therapy (CPT).
  Cognitive Processing Therapy: CPT is a cognitive therapy based on information processing theory and includes components which help the client to (a) access her or his memory of the event, (b) identify and experience her or his emotions until they have been extinguished, and (c) identify and challenge beliefs about the event itself and beliefs about self and the world which have been altered because of the rape.
- Present Centered Therapy (PCT): Participants receive 12 biweekly sessions of Present Centered Therapy (PCT).
  Present-Centered Therapy: PCT consists of general support and education focused on current issues in the patient's life. It emphasizes the focus on the individual's current life, and conceptualizes the problems addressed as manifestations of PTSD that, in some cases, may have been present for long periods of time. Emphasis is on problem solving and improving relationships. Connections are made between current problems and PTSD symptoms. PCT provides the emotional support for the trauma patient that is thought to help in recovery and helps the victim gain a better understanding of the nature of the patient's problems and connection with PTSD.
Period: Overall Study
Arm/Group | Cognitive Processing Therapy (CPT) | Present Centered Therapy (PCT)
Started | 72 | 57
Completed | 44 | 44
Not Completed | 28 | 13

BASELINE CHARACTERISTICS:
Population: Numbers differ from enrollment due to participants excluded from data analysis for poor psychotherapeutic fidelity.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 52 | 34 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.5) | 48.4 (10.7) | 46.1 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 34 | 85
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 30 | 73
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 52 | 34 | 86
PTSD Checklist [Mean (Standard Deviation); unit: units on a scale] — The PCL is a 17-item self-report measure that is commonly used in clinical and research settings. All 17 items are summed to compute a total score of PTSD symptomatology. Scores for the PCL range from 17-85, with 85 indicating severe PTSD symptomatology.The PCL has strong psychometric properties and mirrors the symptomatology of the DSM.
  units on a scale | 65.96 (10.63) | 65.21 (13.25) | 65.65 (11.69)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Checklist (PCL)
Description: The PCL is a 17-item self-report measure that is commonly used in clinical and research settings. All 17 items are summed to compute a total score of PTSD symptomatology. Scores for the PCL range from 17-85, with 85 indicating severe PTSD symptomatology. The PCL has strong psychometric properties and mirrors the symptomatology of the DSM.
Time Frame: Baseline assessment and then 4, follow-up assessments: at treatment completion, 2-month post treatment, 4-month post treatment, and 6-month post treatment
Population: Numbers differ from enrollment due to participants excluded from data analysis for poor psychotherapeutic fidelity.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Processing Therapy (CPT) | Present Centered Therapy (PCT)
Number analyzed (Participants) | 52 | 34
units on a scale
  Baseline | 65.53 (1.67) | 65.40 (2.00)
  Posttreatment (12 Sessions) | 51.39 (2.02) | 57.89 (2.18)
  2-month follow-up | 52.71 (1.98) | 59.35 (2.24)
  4-month follow-up | 54.98 (1.99) | 55.22 (2.15)
  6-month follow-up | 50.52 (1.97) | 56.22 (2.17)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 8/72 | 5/57
Other Adverse Events (participants affected / at risk) | 0/72 | 0/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=72) | Arm 2 (N=57)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) — Some participants reported increased anxiety following participation in talk therapy.
Hospitalization (Psychiatric disorders) | 5 (5) | 3 (3) — Some participants were hospitalized with symptoms related to pain, fatigue, "blacking out," and/or interpersonal violence. None of these were found to be related to their participation in talk therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes